CLINICAL TRIAL: NCT03624127
Title: A Multi-Center, Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: Effectiveness and Safety of BMS-986165 Compared to Placebo and Active Comparator in Participants With Psoriasis
Acronym: POETYK-PSO-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-046; 2018-001926-25 (EudraCT Number)
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib; apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Apremilast (Active Comparator)
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: BMS-986165
Other: Placebo — Specified dose on specified days
  Arms: Placebo
Drug: Apremilast — Specified dose on specified days
  Arms: Apremilast

SUMMARY:
The purpose of this study is to investigate the experimental medication BMS-986165 compared to placebo and a currently available treatment in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Plaque psoriasis for at least 6 months
* Moderate to severe disease
* Candidate for phototherapy or systemic therapy

Exclusion Criteria:

* Other forms of psoriasis
* History of recent infection
* Prior exposure to BMS-986165 or active comparator

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (162):
- United States (67):
  - Achieve Clinical Research, Birmingham, Alabama
  - Coastal Clinical Research - Mobile, Mobile, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Synexus - Tucson, Tucson, Arizona
  - Hull Dermatology, Rogers, Arkansas
  - First OC Dermatology & Belle-Aimee Skincare Clinic Fountain Valley, Fountain Valley, California
  - University California at Irvine Dermatology Clinical Research Center, Irvine, California
  - Keck School of Medicine, Los Angeles, California
  - Dream Team Clinical Research, Pomona, California
  - University Dermatology Group, San Diego, California
  - Unison Clinical Trials, Sherman Oaks, California
  - New England Research Associates, Bridgeport, Connecticut
  - Precision Clinical Research, Davie, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - LCC Medical Research, Miami, Florida
  - International Dermatology Research, Miami, Florida
  - Well Pharma Medical Research, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Renstar Medical Research, Ocala, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Hamilton Dermatology, Alpharetta, Georgia
  - Healthcare Research Network - Flossmoor, Flossmoor, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - The Dermatology Center, New Albany, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Kansas City Dermatology, Overland Park, Kansas
  - Dermatology Specialists Research-Kentucky, Louisville, Kentucky
  - Clinical Trials of America - Monroe, Monroe, Louisiana
  - Etre Cosmetic Dermatology and Laser Center, New Orleans, Louisiana
  - ActivMed Practices and Research - Beverly, Beverly, Massachusetts
  - DermCare Experts, Quincy, Massachusetts
  - David Fivenson MD Dermatology, Ann Arbor, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Associated Skin Care Specialists - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hassman Research Institute, Berlin, New Jersey
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Mount Sinai - Queens, New York, New York
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Duke University Health System - Duke Clinic, Durham, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Synexus - Columbus, Columbus, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Synexus Clinical Research - Anderson, Anderson, South Carolina
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Interspond - Stones River Dermatology - Murfreesboro Office, Murfreesboro, Tennessee
  - Westlake Dermatology - Westlake, Austin, Texas
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Austin Institute for Clinical Research - Pflugerville, Pflugerville, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Interspond - Acclaim Dermatology, Sugar Land, Texas
  - Center for Clinical Studies - Webster, Webster, Texas
  - Dermatology Associates of Seattle, Seattle, Washington
  - Eastern Washington Dermatology, Walla Walla, Washington
- Canada (13):
  - Kirk Barber Research, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Wiseman Dermatology Research, Winnipeg, Manitoba
  - The Guenther Dermatology Research Centre, London, Ontario
  - Office of Dr. Arnon Moshe Katz, Newmarket, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Institute of Cosmetic and Laser Surgery, Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology - Richmond Hill, Richmond Hill, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Docteur David Gratton Dermatologue, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Québec, Quebec
- China (3):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Wuhan, Hubei
  - Local Institution, Hangzhou, Zhejiang
- Germany (2):
  - Charite Universitatsmedizin Berlin, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
- Japan (26):
  - Local Institution - 0165, Nagoya, Aichi-ken
  - Local Institution - 0181, Toon-Shi, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Local Institution - 0182, Isehara, Kanagawa
  - Local Institution - 0169, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nakoku, Kochi
  - University Hospital - Kyoto Preferctural University of Medicine, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Local Institution - 0166, Matsumoto, Nagano
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Teikyo University Hospital, Itabashi-Ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Local Institution - 0188, Shinagawa, Tokyo
  - Local Institution - 0108, Shinjuku, Tokyo
  - Local Institution - 0175, Shinjuku-Ku, Tokyo
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Local Institution - 0167, Osaka
  - Local Institution - 0160, Osaka
- Poland (16):
  - Local Institution - 0191, Warsaw, Masovian Voivodeship
  - Local Institution - 0201, Bialystok
  - Local Institution - 0144, Gdynia
  - Synexus - Katowice, Katowice
  - Local Institution - 0079, Krak
  - Centrum Terapii Wspolczesnej, Lodz
  - Centrum Medyczne All-Med, Lodz
  - Miejski Szpital Zespolony w Olsztynie, Olsztyn
  - DermoDent - Centrum Medyczne Czajkowscy, Osielsko
  - Solumed Centrum Medyczne, Poznan
  - Local Institution - 0200, Poznan
  - Clinical Research Group, Warsaw
  - Center for Clinical Studies - Texas Medical Center, Wroclaw
  - Lukasz Matusiak 4health, Wroclaw
  - dermMedica Sp. z o.o., Wroclaw
  - Local Institution - 0203, Wroclaw
- Russia (13):
  - Azbuka Zdorovya Medical Center, Kazan'
  - Local Institution - 0172, Krasnodar
  - Local Institution - 0140, Moscow
  - Clinical Medical Center of Moscow State Medico-Stomatological University named after AI Evdokimov, Moscow
  - State budgetary institution of Ryazan region - Regional Clinical Skin and Venereal Dispensary, Ryazan
  - Clinic of Skin Diseases of Pierre Wolkenstein, Saint Petersburg
  - Polyclinic of Private Security Personnel, Saint Petersburg
  - Saint-Petersburg SBHI Dermatological and Venereological Dispensary No. 10 - Clinic of Dermatology, Saint Petersburg
  - Ars Vitae Multidisciplinary Medical Center, Saint Petersburg
  - Klinika Kozhnykh I Venericheskikh Bolezney, Saratov
  - Smolensk State Medical University, Smolensk
  - MUZ Clinical Hospital of Emergency Medical Care n.a. N.V. Soloviev, Yaroslavl
  - Local Institution - 0131, Yekaterinburg
- South Korea (6):
  - Local Institution, Busan
  - Local Institution - 0187, Hwaseong-si
  - Local Institution, Hwaseong-si
  - Local Institution, Incheon
  - Local Institution, Seongnam-si
  - Local Institution, Seoul
- Spain (7):
  - Local Institution - 0121, Alcorcón
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Cruces, Barakaldo
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Local Institution - 0097, Valencia
- Taiwan (2):
  - Local Institution, Kaohsiung City
  - Local Institution, Taipei
- United Kingdom (7):
  - MAC Clinical Research - Blackpool, Lancashire
  - Synexus - Merseyside Clinical Research Centre, Liverpool
  - Guys and Saint Thomas NHS Foundation Trust, London
  - Synexus - Manchester Clinical Research Centre, Manchester
  - Salford Royal NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - MAC Clinical Research - Liverpool, Prescot

REFERENCES:
- [Derived] Armstrong AW, Warren RB, Sofen H, Spelman L, Linaberry M, Becker B, Jou YM, Daamen C, Kimball AB. Deucravacitinib in Plaque Psoriasis After Inadequate Response to Apremilast: Phase 3 POETYK Analysis. Dermatol Ther (Heidelb). 2025 Dec 5. doi: 10.1007/s13555-025-01606-9. Online ahead of print. PMID 41350512
- [Derived] Armstrong AW, Kircik L, Stein Gold L, Strober B, De Oliveira CHMC, Vaile J, Jou YM, Daamen C, Scharnitz T, Lebwohl M. Deucravacitinib: Laboratory Parameters Across Phase 3 Plaque Psoriasis Trials. Dermatol Ther (Heidelb). 2025 Apr;15(4):1025-1035. doi: 10.1007/s13555-025-01362-w. Epub 2025 Mar 20. PMID 40113724
- [Derived] Morita A, Imafuku S, Tada Y, Okubo Y, Habiro K, Tsuritani K, Banerjee S, Hoyt K, Kisa RM, Ohtsuki M. Deucravacitinib in plaque psoriasis: Safety and efficacy through 3 years in Japanese patients in the phase 3 POETYK PSO-1, PSO-4, and LTE trials. J Dermatol. 2025 May;52(5):761-772. doi: 10.1111/1346-8138.17685. Epub 2025 Mar 11. PMID 40066907
- [Derived] Armstrong AW, Lebwohl M, Warren RB, Sofen H, Imafuku S, Ohtsuki M, Spelman L, Passeron T, Papp KA, Kisa RM, Vaile J, Berger V, Vritzali E, Hoyt K, Colombo MJ, Scotto J, Banerjee S, Strober B, Thaci D, Blauvelt A. Safety and Efficacy of Deucravacitinib in Moderate to Severe Plaque Psoriasis for Up to 3 Years: An Open-Label Extension of Randomized Clinical Trials. JAMA Dermatol. 2025 Jan 1;161(1):56-66. doi: 10.1001/jamadermatol.2024.4688. PMID 39602111
- [Derived] Armstrong AW, Augustin M, Beaumont JL, Pham TP, Hudgens S, Gordon KB, Zhuo J, Becker B, Zhong Y, Kisa RM, Banerjee S, Papp KA. Deucravacitinib Improves Patient-Reported Outcomes in Patients with Moderate to Severe Psoriasis: Results from the Phase 3 Randomized POETYK PSO-1 and PSO-2 Trials. Dermatol Ther (Heidelb). 2024 Aug;14(8):2235-2248. doi: 10.1007/s13555-024-01224-x. Epub 2024 Jul 30. PMID 39080153
- [Derived] Armstrong AW, Park SH, Patel V, Nicolas P, Wang WJ, Colombo MJ, Chirikov V. Cumulative Benefit Over 52 Weeks With Deucravacitinib Versus Apremilast in Moderate to Severe Plaque Psoriasis: POETYK PSO-1 Post Hoc Analysis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1891-1899. doi: 10.1007/s13555-024-01201-4. Epub 2024 Jun 22. PMID 38907877
- [Derived] Armstrong AW, Gooderham M, Warren RB, Papp KA, Strober B, Thaci D, Morita A, Szepietowski JC, Imafuku S, Colston E, Throup J, Kundu S, Schoenfeld S, Linaberry M, Banerjee S, Blauvelt A. Treatment of plaque psoriasis with deucravacitinib (POETYK PSO-1 study): a plain language summary. Immunotherapy. 2023 Aug;15(12):963-973. doi: 10.2217/imt-2023-0061. Epub 2023 May 7. PMID 37150952
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-986165: BMS-986165 6 mg daily (QD) week 0 - week 52. At week 16, participants were switched in blinded manner from placebo. At week 24, participants who did not achieve PASI 50 were switched in a blinded manner from Apremilast
- Placebo: Participants received placebo week 0 - week 16 and then switched in a blinded manner to BMS-986165 6 mg daily (QD) through week 52
- Apremilast: Apremilast titrated from 10 mg daily (QD) to 30 mg twice a day (BID) over the first 5 days of dosing, continuing through week 24. At week 24, participants who achieved Psoriasis Area and Severity Index (PASI) 50 continued with regimen in a blinded manner and participants who did not achieve PASI 50 were switched in a blinded manner to BMS-986165 6 mg QD through week 52
Period: Pre-treatment
Arm/Group | BMS-986165 | Placebo | Apremilast
Started (Started = Randomized) | 332 | 166 | 168
Completed (Completed = Entered treatment period) | 332 | 165 | 168
Not Completed | 0 | 1 | 0
Not completed — Participant discontinued from study prior to treatment due to incorrect randomization | 0 | 1 | 0
Period: Treatment Week 0 - Week 16
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 332 | 165 | 168
Completed | 307 | 145 | 145
Not Completed | 25 | 20 | 23
Not completed — Adverse Event | 5 | 7 | 10
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Lost to Follow-up | 7 | 2 | 4
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 3
Not completed — Other reasons | 8 | 5 | 3
Period: Treatment Week 16 - Week 24
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 452 | 0 | 145
Completed | 442 | 0 | 141
Not Completed | 10 | 0 | 4
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Other reasons | 3 | 0 | 0
Period: Treatment Week 24 - Week 52
Arm/Group | BMS-986165 | Placebo | Apremilast
Started | 496 | 0 | 87
Completed | 444 | 0 | 83
Not Completed | 52 | 0 | 4
Not completed — Adverse Event | 8 | 0 | 1
Not completed — Lack of Efficacy | 6 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Site terminated by sponsor | 2 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0
Not completed — Other reasons | 19 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986165 | Placebo | Apremilast | Total
Number analyzed (Participants) | 332 | 166 | 168 | 666
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (13.71) | 47.9 (13.98) | 44.7 (12.06) | 46.1 (13.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 53 | 58 | 213
  Male | 230 | 113 | 110 | 453
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 26 | 30 | 106
  Not Hispanic or Latino | 282 | 140 | 138 | 560
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 267 | 128 | 139 | 534
  Black or African American | 2 | 3 | 1 | 6
  Asian | 59 | 34 | 28 | 121
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Other | 4 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Static Physician's Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (sPGA 0/1)
Description: The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. The higher sPGA score denotes to more severe disease activity (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; Severe = 4). sPGA 0/1 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as 0 or 1 with at least 2-point improvement from baseline using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 16 or who have missing week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants in BMS-986165 and Placebo arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 332 | 166
Participants | 178 | 12
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 18.71, 95% CI 2-sided [9.51 to 36.81]

2. Primary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (PASI 75)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the response as a number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 16 or who have missing week 16 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline and Week 16
Population: All randomized participants in BMS-986165 and Placebo arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 332 | 166
Participants | 194 | 21
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 11.09, 95% CI 2-sided [6.49 to 18.95]

3. Secondary Outcome: The Number of Participants Who Achieve a 90% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score at Week 16 (PASI 90)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the response as a number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 16 or who have missing week 16 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline and Week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 332 | 166 | 168
Participants | 118 | 7 | 33
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 16.15, 95% CI 2-sided [6.91 to 37.72]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.40, 95% CI 2-sided [1.51 to 3.60]

4. Secondary Outcome: The Number of Participants Who Achieve a 100% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (PASI 100)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 100 is the response as a number of participants who experience at least a 100% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 16 or who have missing week 16 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline and Week 16
Population: Pre-specified for data to be collected only in all randomized from BMS-986165 and Placebo Arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 332 | 166
Participants | 47 | 1
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 31.30, 95% CI 2-sided [4.09 to 239.36]

5. Secondary Outcome: The Number of Participants With a Static Physician's Global Assessment Score of 0 at Week 16 (sPGA 0)
Description: The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. The higher sPGA score denotes to more severe disease activity (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; 4 = Severe). sPGA 0 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as 0 using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 16 or who have missing week 16 endpoint data for any reason.
Time Frame: Week 16
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 332 | 166 | 168
Participants | 58 | 1 | 8
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.52, 95% CI 2-sided [2.07 to 9.84]
Statistical Analysis 2: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 39.54, 95% CI 2-sided [5.29 to 295.75]

6. Secondary Outcome: Change From Baseline in Psoriasis Symptoms and Signs Diary (PSSD) Symptom Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 16
Description: PSSD is an 11-item participant-reported instrument that assesses severity of symptoms and participant-observed signs commonly associated in plaque psoriasis. PSSD assesses severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 participants-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding) using 0-10 numerical ratings. The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). A symptom score will be derived by averaging the 5 questions and multiplying by 10. A sign score will be derived by averaging the 6 questions and multiplying by 10. A total PSSD score with range 0-100 will be derived from taking the average of the symptom and sign scores, where 0 representing the least severe symptom/sign and 100 the most severe. A mBOCF approach will be used for missing data.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline and Week 16
Population: Pre-specified for data to be collected only in all responders from BMS-986165 and Apremilast Arms
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 306 | 158
Score on a scale | -29.4 (24.43) | -22.8 (23.40)
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Mean Difference = -8.8, 95% CI 2-sided [-12.8 to -4.9], Standard Error of Mean 2.00

7. Secondary Outcome: Psoriasis Symptoms and Signs Diary (PSSD) Symptom Score 0 at Week 16
Description: PSSD with a 24-hour recall period is an 11-item participant-reported instrument that assesses severity of symptoms and participant-observed signs commonly associated in plaque psoriasis. PSSD assesses severity of 5 symptoms (itch, pain, stinging, burning, skin tightness) and 6 participants-observed signs (skin dryness, cracking, scaling, shedding or flaking, redness, bleeding) using 0-10 numerical ratings. The severity of each item is rated on an 11-point numeric rating scale ranging from 0 (absent) to 10 (worst imaginable). PSSD 0 is the response as a number of participants who experience a PSSD symptom score that is derived from the average of the scores and determines psoriasis severity as 0 among participants with a baseline PSSD symptom score >= 1.
Time Frame: Week 16
Population: All Responders with a baseline PSSD symptom score >= 1
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 305 | 149 | 158
Participants | 24 | 1 | 7
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 13.67, 95% CI 2-sided [1.77 to 105.50]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.1702, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.76 to 4.42]

8. Secondary Outcome: The Number of Participants With a Dermatology Life Quality Index (DLQI) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Placebo at Week 16 (DLQI 0/1)
Description: DLQI is a participant-reported quality of life index which consists of 10 questions concerning symptoms and feelings, daily activities, leisure, work, school, personal relationships, and treatment during the last week before questionnaire. Each question is scored on a scale of 0 to 3 by a tick box (0 = "not at all"; 1 = "a little"; 2 = "a lot"; or 3 = "very much"). The scores are summed, giving a range from 0 (no impairment of life quality) to 30 (maximum impairment). DLQI 0/1 is the response as a number of participants who experience DLQI score of 0 or 1 among participants with a baseline DLQI score >=2.
Time Frame: Week 16
Population: Pre-specified for data to be collected only in all responders with a baseline DLQI score >=2 from BMS-986165 and Placebo Arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 322 | 160
Participants | 132 | 17
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.04, 95% CI 2-sided [3.46 to 10.53]

9. Secondary Outcome: Number of Participants With a Physician's Global Assessment-Fingernails (PGA-F) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Placebo at Week 16
Description: PGA-F overall condition of the fingernails is rated on a 5-point scale (0 = clear; 1 = minimal; 2 = mild; 3 = moderate; and 4 = severe). PGA-F 0/1 is the response as a number of participants with a PGA-F score of 0 or 1 with at least a 2-point improvement from baseline among participants with a baseline PGA-F score >=3.
Time Frame: Week 16
Population: Pre-specified for data to be collected only in all responders with a baseline PGA-F score >=3 from BMS-986165 and Placebo Arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo
Number analyzed (Participants) | 43 | 34
Participants | 9 | 3
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p = 0.1049, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.84, 95% CI 2-sided [0.73 to 10.96]

10. Secondary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 16 (PASI 75)
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: All randomized participants in BMS-986165 and Apremilast arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 168
Participants | 194 | 59
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.78 to 3.91]

11. Secondary Outcome: The Number of Participants With a Static Physician's Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Apremilast at Week 16 (sPGA 0/1)
Description: as for outcome 1
Time Frame: Week 16
Population: All randomized participants in BMS-986165 and Apremilast arms
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 168
Participants | 178 | 54
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.70 to 3.78]

12. Secondary Outcome: The Number of Participants With a Scalp Specific Physician's Global Assessment (Ss-PGA) Score 0 or 1 at Week 16 (Ss-PGA 0/1)
Description: ss-PGA is a 5-point scale that evaluates scalp lesions in terms of clinical signs of redness, thickness, and scaliness. The higher ss-PGA score denotes to more severe disease activity (0 = absence of disease; 1 = very mild disease; 2 = mild disease; 3 = moderate disease; 4 = severe disease). ss-PGA 0/1 is the response as a number of participants who experience a ss-PGA score that determines scalp lesions severity as 0 or 1 with at least a 2-point improvement from baseline among participants with a baseline ss-PGA score >=3.
Time Frame: Week 16
Population: All responders with a baseline ss-PGA score >=3
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Placebo | Apremilast
Number analyzed (Participants) | 209 | 121 | 110
Participants | 147 | 21 | 43
Statistical Analysis 1: Comparison: BMS-986165 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 11.92, 95% CI 2-sided [6.69 to 21.25]
Statistical Analysis 2: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.65, 95% CI 2-sided [2.21 to 6.04]

13. Secondary Outcome: The Number of Participants With a Static Physician's Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Apremilast at Week 24 (sPGA 0/1)
Description: The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. The higher sPGA score denotes to more severe disease activity (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; Severe = 4). sPGA 0/1 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as 0 or 1 with at least 2-point improvement from baseline using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 24 or who have missing week 24 endpoint data for any reason.
Time Frame: Week 24
Population: Pre-specified for data to be collected in all randomized who received BMS-986165 only and Apremilast
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 168
Participants | 195 | 52
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.23, 95% CI 2-sided [2.16 to 4.83]

14. Secondary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 24 (PASI 75)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the response as a number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 24 or who have missing week 24 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline and Week 24
Population: Pre-specified for data to be collected in all randomized who received BMS-986165 only and Apremilast
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 168
Participants | 230 | 64
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.76, 95% CI 2-sided [2.53 to 5.60]

15. Secondary Outcome: The Number of Participants Who Achieve a 90% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 24 (PASI 90)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the response as a number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 24 or who have missing week 24 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline and Week 24
Population: Pre-specified for data to be collected in all randomized who received BMS-986165 only and Apremilast
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 168
Participants | 140 | 37
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.71 to 4.05]

16. Secondary Outcome: The Number of Participants With a Static Physician's Global Assessment (sPGA) Score of 0 or 1 in Participants Receiving BMS-986165 Compared to Apremilast at Week 52 and at Week 24 (sPGA 0/1)
Description: The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. The average of the 3 scales, which is rounded to the nearest whole number, is the final sPGA score. The higher sPGA score denotes to more severe disease activity (0 = Clear; 1 = Almost clear; 2 = Mild; 3 = Moderate; Severe = 4). sPGA 0/1 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as 0 or 1 with at least 2-point improvement from baseline using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 52 or who have missing week 52 endpoint data for any reason.
Time Frame: Week 52 and Week 24
Population: Pre-specified for data to be collected in all responders treated in BMS-986165 arm and Apremilast arm
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 167
Participants | 151 | 37
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.96 to 4.69]

17. Secondary Outcome: The Number of Participants Who Achieve a 75% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 52 and at Week 24 (PASI 75)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the response as a number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 52, or who have missing week 52 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline, Week 52 and Week 24
Population: Pre-specified for data to be collected in all responders treated in BMS-986165 arm and Apremilast arm
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 167
Participants | 187 | 51
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.11, 95% CI 2-sided [2.06 to 4.69]

18. Secondary Outcome: The Number of Participants Who Achieve a 90% Improvement From Baseline in the Psoriasis Area and Severity Index (PASI) Score in Participants Receiving BMS-986165 Compared to Apremilast at Week 52 and at Week 24 (PASI 90)
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 90 is the response as a number of participants who experience at least a 90% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method that will be used for participants who discontinue treatment or study prior to week 52, or who have missing week 52 endpoint data for any reason.
  Baseline is defined as the measurement at the randomization visit (Week 0).
Time Frame: Baseline, Week 52 and Week 24
Population: Pre-specified for data to be collected in all responders treated in BMS-986165 arm and Apremilast arm
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 | Apremilast
Number analyzed (Participants) | 332 | 167
Participants | 103 | 26
Statistical Analysis 1: Comparison: BMS-986165 vs Apremilast; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.55 to 4.19]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-cause mortality from their first dose to study completion (up to approximately 24 months). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 12 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- BMS-986165 Week 0 up to Week 16: BMS-986165 6 mg daily (QD) week 0 - week 16
- Placebo Week 0 up to Week 16: Participants received placebo week 0 - week 16
- Apremilast Week 0 up to Week 16: Apremilast titrated from 10 mg daily (QD) to 30 mg twice a day (BID) over the first 5 days of dosing week 0 - week 16
- BMS-986165 Week 0 up to Week 52: BMS-986165 6 mg daily (QD) week 0 - week 52
- Placebo Week 0 up to Week 52: Participants received placebo week 0 - week 52
- Apremilast Week 0 up to Week 52: Apremilast titrated from 10 mg daily (QD) to 30 mg twice a day (BID) over the first 5 days of dosing week 0 - week 52
Arm/Group | BMS-986165 Week 0 up to Week 16 | Placebo Week 0 up to Week 16 | Apremilast Week 0 up to Week 16 | BMS-986165 Week 0 up to Week 52 | Placebo Week 0 up to Week 52 | Apremilast Week 0 up to Week 52
All-Cause Mortality (participants affected / at risk) | 0/332 | 1/166 | 0/168 | 0/531 | 1/166 | 0/168
Serious Adverse Events (participants affected / at risk) | 7/332 | 9/165 | 4/168 | 31/531 | 9/165 | 6/168
Other Adverse Events (participants affected / at risk) | 76/332 | 24/165 | 60/168 | 197/531 | 24/165 | 80/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 Week 0 up to Week 16 (N=332) | Placebo Week 0 up to Week 16 (N=165) | Apremilast Week 0 up to Week 16 (N=168) | BMS-986165 Week 0 up to Week 52 (N=531) | Placebo Week 0 up to Week 52 (N=165) | Apremilast Week 0 up to Week 52 (N=168)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Hernia perforation (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 Week 0 up to Week 16 (N=332) | Placebo Week 0 up to Week 16 (N=165) | Apremilast Week 0 up to Week 16 (N=168) | BMS-986165 Week 0 up to Week 52 (N=531) | Placebo Week 0 up to Week 52 (N=165) | Apremilast Week 0 up to Week 52 (N=168)
Diarrhoea (Gastrointestinal disorders) | 13 | 6 | 17 | 30 | 6 | 19
Nausea (Gastrointestinal disorders) | 7 | 4 | 19 | 7 | 4 | 21
Nasopharyngitis (Infections and infestations) | 21 | 7 | 14 | 96 | 7 | 26
Upper respiratory tract infection (Infections and infestations) | 21 | 6 | 3 | 50 | 6 | 6
Headache (Nervous system disorders) | 16 | 5 | 17 | 35 | 5 | 23
Hypertension (Vascular disorders) | 6 | 0 | 6 | 14 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03624127/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03624127/SAP_001.pdf